CLINICAL TRIAL: NCT00283543
Title: A Phase II Study of Radiation With Concomitant and Then Sequential Temozolomide in Patients With Newly Diagnosed Supratentorial Malignant Glioma Who Have Undergone Surgery With Gliadel Wafer Insertion
Brief Title: Radiation With Concomitant and Then Sequential Temozolomide in Malignant Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kentuckiana Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1068016; 128-02
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Newly Diagnosed Supratentorial Malignant Glioma
Keywords: Glioma; Gliadel Wafer
MeSH Terms: conditions — Glioma | interventions — Carmustine; Temozolomide

INTERVENTIONS:
Drug: Gliadel Wafer
Drug: Temozolomide
Procedure: Limited field radiation

SUMMARY:
To determine the safety and efficacy of Gliadel 3.85% wafers plus surgery and radiation with Temozolomide

DETAILED DESCRIPTION:
A phase II study of radiation with concomitant and then sequential Temozolomide in patients with newly diagnosed supratentorial malignant glioma who have undergone surgery with Gliadel wafer insertion. To determine the safety and efficacy of Gliadel 3.85% wafers plus surgery and limited field radiation therapy with concomitant Temozolomide followed by Temozolomide alone in patients undergoing initial surgery for newly diagnosed unifocal moderate to high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* MRI showing unilateral supratentorial cerebral tumor
* surgical tx within 4 weeks of baseline MRI
* KPS 60% or higher
* moderate to high grade malignant glioma

Exclusion Criteria:

* prior cytoreductive surgery for moderate or high grade glioma
* prior CNS radiotherapy
* prior chemo for this glioma
* more than one focus of tumor or tumor crossing the midline per MRI
* life expectancy less than 12 months
* sensitivity to temozolomide, nitrosoureas, or Gliadel wafer

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-09; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and efficacy of Gliadel 3.85% wafers

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, Study Director — Kentuckiana Cancer Institute
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States